CLINICAL TRIAL: NCT04607707
Title: Satisfaction and Treatment Adherence in Women With Vulvovaginal Atrophy: A Cross-sectional Study (CRETA Study)
Brief Title: Women's Satisfaction and Adherence to Vulvovaginal Atrophy Treatments
Acronym: CRETA
Status: Completed | Type: Observational
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Other Study IDs: CRETA
Record Dates: First submitted 2020-09-22; First posted 2020-10-29 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Vulvovaginal Atrophy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postmenopausal Women: Participants who sign an informed consent will be asked to complete study questionnaires at a single visit that coincides with a normal healthcare visit. No other study procedures will be performed.

SUMMARY:
The primary objective of this study is to describe and assess participants' satisfaction with current vulvovaginal atrophy (VVA) treatment.

DETAILED DESCRIPTION:
This study is designed as a multicenter, cross-sectional, descriptive, observational study.

ELIGIBILITY:
Inclusion Criteria:

* Women with natural menopause established for at least one year.
* Absence of menstruation for at least one year.
* Mild, moderate or severe VVA diagnosis.
* Currently under treatment with either Ospemifene, Local Oestrogen Therapy or moisturizers for at least 3 months in accordance with the approved SmPC and/or Patient Leaflet
* Patients providing writing informed consent for participating in the study.

Exclusion Criteria:

* Women who have never been previously treated for VVA
* Women who have discontinued their VVA treatment due to a contraindication in the study group drug.
* Patients using more than one VVA treatment at a time (except for lubricants).
* Breastfeeding, pregnancy or under any kind of systemic hormonal treatment that causes amenorrhea.
* Local phytotherapy for VVA.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Post-menopausal women visiting gynecologists at Spanish public and private centers.
Sampling Method: Non-Probability Sample
Enrollment: 831 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Perception of Patient Satisfaction with Their Current Vulvovaginal Atrophy (VVA) Treatment by means of a questionnaire | Day 0
  The results will be determined by an evaluation the patient's selection of answers to 32 questions designed to determine the patient's use of, compliance with, and satisfaction with treatments for vulvovaginal atrophy. The questions have answers on a 5-point scale with the lowest score for dissatisfaction and the highest score for satisfaction
Perception of Patient Satisfaction with Long-term VVA Treatment of Vulvovaginal Atrophy by Means of a Questionnaire | Day 0
  The results will be determined by an evaluation the patient's selection of answers to 32 questions designed to determine the patient's use of, compliance with, and satisfaction with treatments for vulvovaginal atrophy. The questions have answers on a 5-point scale with the lowest score for dissatisfaction and the highest score for satisfaction

SECONDARY OUTCOMES:
Factors that the Patient Identifies as Advantages of VVA Treatment by Means of a Questionnaire | Day 0
  The results will be determined by an evaluation the patient's selection of answers to 32 questions designed to determine the patient's use of, compliance with, and satisfaction with treatments for vulvovaginal atrophy. The questions have answers on a 5-point scale with the lowest score for dissatisfaction and the highest score for satisfaction
Factors that the Patient Identifies as Disadvantages of VVA Treatment by Means of a Questionnaire | Day 0
  The results will be determined by an evaluation the patient's selection of answers to 32 questions designed to determine the patient's use of, compliance with, and satisfaction with treatments for vulvovaginal atrophy. The questions have answers on a 5-point scale with the lowest score for dissatisfaction and the highest score for satisfaction
Preferred Route of Administration and Treatment Schedule for VVA Determined by a Questionnaire | Day 0
  The results will be determined by an evaluation the patient's selection of answers to 32 questions designed to determine the patient's use of, compliance with, and satisfaction with treatments for vulvovaginal atrophy. The questions have answers on a 5-point scale with the lowest score for dissatisfaction and the highest score for satisfaction
Other Factors that Affect Adherence to VVA Treatment in the Patient´s Opinion as Determined by a Questionnaire | Day 0
  The results will be determined by an evaluation the patient's selection of answers to 32 questions designed to determine the patient's use of, compliance with, and satisfaction with treatments for vulvovaginal atrophy. The questions have answers on a 5-point scale with the lowest score for dissatisfaction and the highest score for satisfaction
Treatment Most Rejected by Patients According to the Opinion of the Healthcare Professional (HCP) | Day 0
Preferred Route of Administration and Treatment Schedule in the Opinion of the HCP | Day 0
Factors the HCP Identifies as Advantages of VVA Treatment by Means of a Questionnaire | Day 0
  The results will be determined by an evaluation the HCP's selection of answers to 32 questions designed to determine the patient's use of, compliance with, and satisfaction with treatments for vulvovaginal atrophy. The questions have answers on a 5-point scale with the lowest score for dissatisfaction and the highest score for satisfaction
Factors the HCP Identifies as Disadvantages of VVA Treatment by Means of a Questionnaire | Day 0
  The results will be determined by an evaluation the HCP's selection of answers to 32 questions designed to determine the patient's use of, compliance with, and satisfaction with treatments for vulvovaginal atrophy. The questions have answers on a 5-point scale with the lowest score for dissatisfaction and the highest score for satisfaction
HCP's Perception of Treatment Duration for Each Type of VVA Treatment | Day 0
Other Factors that Influence Adherence According to the HCP Determined by Means of a Questionnaire | Day 0
  The results will be determined by an evaluation the HCP's selection of answers to questions designed to determine the patient's use of, compliance with, and satisfaction with treatments for vulvovaginal atrophy. The questions have answers on a 5-point scale with the lowest score for dissatisfaction and the highest score for satisfaction
HCP´s Perception about Patient Non-compliance to Each of the VVA Treatments | Day 0
Treatment Duration for Each Type of VVA Treatment According to the HCP and the Patient | Day 0
Patients' Preferred Treatment, Route of Administration and Treatment Schedule According to the HCP | Day 0
Factors that According to the HCP and the Patient Influence the Patient's Decision to Discontinue Treatment | Day 0
Factors Positively Affecting the Patient's Adherence to Each Treatment According to the HCP and Patient | Day 0
VVA Acknowledgement by the Patient | Day 0
VVA Symptoms Acknowledged by the Patient | Day 0
Satisfaction with Current VVA Treatment by means of a Questionnaire | Day 0
  The results will be determined by an evaluation the patient's selection of answers to 32 questions designed to determine the patient's use of, compliance with, and satisfaction with treatments for vulvovaginal atrophy. The questions have answers on a 5-point scale with the lowest score for dissatisfaction and the highest score for satisfaction
Acknowledgement of the Advantages and Disadvantages of Treatment for VVA | Day 0
Patient's Level of Compliance to the Treatment Scheme Prescribed by the HCP by Means of a Questionnaire | Day 0
  The results will be determined by an evaluation the patient's selection of answers to 32 questions designed to determine the patient's use of, compliance with, and satisfaction with treatments for vulvovaginal atrophy. The questions have answers on a 5-point scale with the lowest score for dissatisfaction and the highest score for satisfaction
Importance Given by the Patient to Comply with the Treatment for VVA | Day 0
Patient Compliance with HCP instructions Regarding the Treatment Dosage by Means of a Questionnaire | Day 0
  The results will be determined by an evaluation the patient's selection of answers to 32 questions designed to determine the patient's use of, compliance with, and satisfaction with treatments for vulvovaginal atrophy. The questions have answers on a 5-point scale with the lowest score for dissatisfaction and the highest score for satisfaction
Reasons for not Following HCP Instructions for Treatment of VVA | Day 0
Importance Patient Gives to Follow the Instructions of her Doctor About the Treatment for VVA | Day 0
Cervantes Quality of Life (QOL) Questionnaire Total Score and Domain Scores | Day 0
Symptoms that Most Benefit from VVA Treatment According to the Patient | Day 0
Time to Improvement in VVA Symptoms According to the Patient | Day 0
Effect of Educational Level, Marital Status, Age, and Geographic Location on Treatment Adherence for VVA | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (3):
- Spain (3):
  - Clínica Teknon, Barcelona
  - Hospital Universitario de Guadalajara, Guadalajara
  - Instituto Palacios, Madrid

REFERENCES:
- [Derived] Palacios S, Sanchez-Borrego R, Suarez Alvarez B, Lugo Salcedo F, Gonzalez Calvo AJ, Quijano Martin JJ, Cancelo MJ, Fasero M. Impact of vulvovaginal atrophy therapies on postmenopausal women's quality of life in the CRETA study measured by the Cervantes scale. Maturitas. 2023 Jun;172:46-51. doi: 10.1016/j.maturitas.2023.03.007. Epub 2023 Mar 30. PMID 37099983